CLINICAL TRIAL: NCT01852669
Title: A Prospective, Randomized, Double Blind, Controlled Study Comparing Extracorporeal Shock Wave Lithotripsy (ESWL) With and Without Simultaneous Adjunct Controlled Inversion Therapy in the Treatment of Lower Pole Caliceal Stone
Brief Title: Adjunct Inversion for Lower Pole Stone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: Lam Wah Ee Hospital (Other)
Responsible Party: Principal Investigator, Shaun Lee Wen Huey, Senior Lecturer, Monash University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LPS001
Record Dates: First submitted 2013-05-02; First posted 2013-05-14 (Estimated); Results first posted 2015-04-20 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inversion, Hydration, ESWL (Experimental): ESWL with hydration and inversion
  Interventions: Procedure: Inversion; Procedure: Shock Wave Lithotripsy; Drug: Hydration
- ESWL, Hydration (Active Comparator): ESWL with hydration
  Interventions: Procedure: Shock Wave Lithotripsy; Drug: Hydration

INTERVENTIONS:
Procedure: Inversion — Patients inverted 30 degree head down in Trendelenburg position
  Arms: Inversion, Hydration, ESWL
Procedure: Shock Wave Lithotripsy — Shock wave lithotripsy
  Other Names: ESWL
Drug: Hydration — Hydration of patient with 0.5L NaCl and 20mg frusemide IV
  Other Names: Frusemide 20mg

SUMMARY:
This is a randomized controlled trial comparing extracorporeal shockwave lithotripsy (ESWL) with and without simultaneous adjunct controlled inversion therapy in the treatment of lower pole caliceal stone.

ELIGIBILITY:
Inclusion Criteria:

1. Solitary lower pole caliceal stone which is > 5 mm and < 20mm
2. Not contraindicated for intravenous urogram (IVU) and subsequent X-rays
3. Patient able to comply strictly with visits/medications
4. Patient willing and agrees to enter study

Exclusion Criteria:

1. Impaired function of the affected kidney
2. Gross hydronephrosis of the affected kidney
3. Associated distal obstruction
4. Multiple stones
5. Stone more than 2 cm in size
6. Diverticular stone
7. Patients who are contraindicated for extracorporeal shockwave lithotripsy e.g.: Pregnancy
8. Patients who are unable to tolerate the procedure
9. Significant cardiac condition that does not allow the administration of force hydration or inversion.
10. Uncontrolled hypertension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2002-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liong Men Long, MBBS, Principal Investigator — Lam Wah Ee Hospital

REFERENCES:
- [Derived] Leong WS, Liong ML, Liong YV, Wu DB, Lee SW. Does simultaneous inversion during extracorporeal shock wave lithotripsy improve stone clearance: a long-term, prospective, single-blind, randomized controlled study. Urology. 2014 Jan;83(1):40-4. doi: 10.1016/j.urology.2013.08.004. Epub 2013 Sep 14. PMID 24044912

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inversion, Hydration, ESWL | ESWL, Hydration
Started | 71 | 69
Completed | 71 | 68 (Randomisation error. Patient has protocol violation which necessitated exclusion from analysis)
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inversion, Hydration, ESWL | ESWL, Hydration | Total
Number analyzed (Participants) | 71 | 68 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (11.1) | 50.9 (12.9) | 49.63 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 51 | 47 | 98

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are Stone Free at 3 Months
Description: To compare the effectiveness of simultaneous adjunct controlled inversion therapy during extracorporeal shockwave lithotripsy (ESWL) to that of ESWL alone in the treatment of lower pole caliceal stone as measured by stone-free rate(SFR)
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Inversion, Hydration, ESWL | ESWL, Hydration
Number analyzed (Participants) | 71 | 68
participants | 54 | 49

ADVERSE EVENTS:
Arm/Group | Inversion, Hydration, ESWL | ESWL, Hydration
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/68
Other Adverse Events (participants affected / at risk) | 1/71 | 2/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inversion, Hydration, ESWL (N=71) | ESWL, Hydration (N=68)
Haematoma (Blood and lymphatic system disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No